CLINICAL TRIAL: NCT06142240
Title: Efficacy of Two Therapeutic Exercise Modalities for Patients With Persistent COVID: Pilot Study
Brief Title: Efficacy of Two Therapeutic Exercise Modalities for Patients With Persistent COVID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Facultat de ciencies de la Salut Universitat Ramon Llull (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-04-02
Record Dates: First submitted 2023-11-08; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Persistent COVID-19
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: Study design: Interventional study. The study will be carried out at the Ricard i Fortuny Social and Health Centre (CSSV RiF) in Vilafranca del Penedès (Barcelona).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- programe at the health centre (Active Comparator): Subjects who are included in the study will perform a therapeutic exercise programme which will have a duration of 8 weeks and 2 sessions per week of 1h duration. Participants assigned to the supervised group will perform the programme at the health centre
  Interventions: Other: exercise programe
- programe at the health home (Experimental): Subjects who are included in the study will perform a therapeutic exercise programme which will have a duration of 8 weeks and 2 sessions per week of 1h duration. Participants assigned to the to the home group will receive telematic supervision (via videoconference).
  Interventions: Other: exercise programe

INTERVENTIONS:
Other: exercise programe — The components of the exercise programe will be: muscle strength training and continuous-variable aerobic training or HIIT with loads between 70-90% of maximum heart rate. The aerobic training will last about 30 minutes and will then be completed with muscle training of the upper and lower limbs with loads determined according to the perception of effort (loads around 50-70%). The sessions will be monitored with pulse oximetry (heart rate and oxygen saturation), perception of fatigue and sensation of suffocation (Borg scale). The intensity of each component of the programme will be individualised according to the conditions of each subject.
  Adherence to the programme will be recorded as successful when participation in the sessions is greater than 80% of the total number of sessions.

SUMMARY:
Symptoms of long-standing sequelae and complications of COVID-19, termed Long COVID19 or persistent COVID, have been reported worldwide. However, the etiology underlying the prolonged or fluctuating symptomatology is limited and there is no uniform and widely accepted definition.Patients describe persistent COVID as a fluctuating disease with variable and persistent symptoms.Most of the effects correspond to clinical symptoms such as fatigue, headache, arthralgias, hyposmia, gustatory sensations, etc. Fatigue is the most common and prolonged symptom of persistent COVID. Knowledge of the pathophysiological mechanisms of fatigue in COVID-19 disease, as well as the therapeutic approach, remains limited due to the relatively recent onset of this pathology. In particular, muscle strength training has been shown to improve muscle function and fatigue, not only during treatment, but also at long-term follow-up.

DETAILED DESCRIPTION:
Objective: To evaluate the effects on the perception of fatigue in patients with persistent COVID, who undergo a supervised and directed therapeutic exercise program in a health center compared to a home therapeutic exercise program.

Methods: Randomized pilot study. Subjects who are included in the study will perform a therapeutic exercise program which will last 8 weeks and 2 sessions per week of 1h duration. The participants assigned to the supervised group will carry out the program at the health center, while the participants assigned to the home group will receive telematic supervision (by videoconference). Both groups will be under the supervision of the assigned physiotherapist.

The components that will form part of the exercise program will be: muscular strength training and continuous-variable aerobic training or HIIT type with loads between 70-90% of maximum heart rate. The main variables are fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients diagnosed with LongCOVID19 or persistent COVID19.
* Agree to participate and sign the informed consent form.

Exclusion Criteria:

* Patients with comorbidities associated with having fatigue (e.g. cancer survivors, severe cardiovascular or respiratory disease prior to persistent COVID).
* Taking medication of drugs that may interfere with the perception of fatigue.
* Patients with mental disorders or cognitive impairment prior to persistent COVID.
* Patients who regularly practice intense sports (>4h/week).
* Any illness that may condition understanding and compliance with the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Fatigue | hour
  this is the main variable of the study. It will be measured using the self-report scale "Fatigue Impact Scale" (FIS) (Fisk et al., 1994), which assesses the perception of functional limitation caused by fatigue in three areas: physical, cognitive and psychosocial. Range 0 (no problem) to 4 (extrem problem)

SECONDARY OUTCOMES:
Exercise capacity | hour
  will be assessed using the six-minute walk test (6MWT). In the 6MWT we will measure the total number of metres the patient is able to walk for 6 minutes. The test will be performed in an indoor corridor of 30m distance, repeated 2 times with a pause of at least 30min between them.

OTHER OUTCOMES:
Pulmonary function | hour
  Spirometry will be measured using an EasyOneTM World Spirometer (ndd Medical Technologies, Zurich, Switzerland).
  * Forced spirometry (FEV1, normal value 70-75% mesure Litres) percentage of the total exhaled volume in the first second
  * Forced vital capacity (FVC, normal value 80% mesure Litres ) It is made up of the sum of total volume, inspiratory reserve volume and expiratory reserve volume.
  The variables will be included in the analysis and will be performed following ATS/ERS recommendations (19).

CONTACTS AND LOCATIONS:
Locations (1):
- CSSV-Rif, Barcelona, Vilafranca Del Penedés, Spain